CLINICAL TRIAL: NCT04978207
Title: COVID-19 Testing and Linkage to Care With Faith-based and Health Agency Partners: A Faithful Response to COVID-19
Brief Title: A Faithful Response to COVID-19 Project
Acronym: FR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Responsible Party: Principal Investigator, Jannette Berkley-Patton, Professor, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB #2038603 KC
Record Dates: First submitted 2021-07-19; First posted 2021-07-27 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: A Multilevel, Tailored COVID-19 Testing Condition; A Nontailored COVID-19 Testing Control Condition
Keywords: African American; Faith-based; COVID-19 testing; Cultural tailoring; Linkage to care; Contact tracing

STUDY DESIGN:
Intervention Model Description: A culturally-religiously tailored COVID-19 testing and linkage to care arm versus a standard COVID-19 education arm in African American churches
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multilevel, religiously-culturally tailored COVID-19 testing and linkage to care (Experimental): Church-based COVID19 promoted with a religiously-culturally tailored Faithful Response COVID19 Toolkit delivered by church health workers (trained in an enhanced communication style) through multilevel church outlets (e.g., sermon guide, responsive reading, church bulletin inserts, automated text messages) and linkage to care delivered by community health workers who also conduct contact tracing; inclusive of 2 church-based COVID-19 testing events at each participating site.
  Interventions: Behavioral: A Faithful Response to COVID-19
- Standard COVID19 information (non-tailored) attention control arm (Active Comparator): Standard COVID-19 information that has not been tailored delivered by trained church health workers via a toolkit; inclusive of 2 church-based COVID19 testing evens at each participating site.
  Interventions: Behavioral: A Faithful Response to COVID-19

INTERVENTIONS:
Behavioral: A Faithful Response to COVID-19 — See previous description

SUMMARY:
This 2-arm clustered, randomized community trial will test a multilevel, COVID-19 testing and linkage to care (eg, health insurance, medical appointments, community resources, contact tracing) intervention against a nontailored, attention-control condition on uptake of COVID-19 testing with adult African American church-affiliated members at 6 months. Contact tracing approval (beliefs and participation contact tracing) and COVID19 prevention behaviors will also be examined. Findings from this study could provide a theory-based, multilevel model for delivering scalable, wide-reaching COVID-19 testing and linkage to care services, including contact tracing, by supporting African American faith leaders with culturally-appropriate, easy-to-use tools and health agency partnerships.

DETAILED DESCRIPTION:
The primary aim of this study is to conduct a two-arm clustered randomized controlled trial to fully test a multilevel, religiously-tailored African American church-based COVID19 testing and linkage to care (LTC) intervention (Tx) vs a nontailored multilevel, attention-control (AC) condition on COVID19 testing uptake (primary outcome) at 6 mos. LTC, contact tracing approval (CTA) and prevention behaviors (exploratory secondary outcomes) will also be examined with participants, adult African American church and community members. Churches will be matched on attendance size and denomination, and randomly assigned to Tx or AC. Previous HIV testing and diabetes prevention studies conducted in African American churches, whereby the Theory of Planned Behavior (TPB) and Socioecological Model will guide intervention design and delivery, will be adapted for this project. Using a community engaged approach, these models provide a theoretically-based, ecologically-expanded TBP framework for intervention delivery through multilevel church outlets to increase reach, dose, and impact. Sixteen churches (45 church members and 15 community members using outreach services per church; N= 960 total) have been project to be required to detect significant increases in testing.

Trained church health workers will deliver the Tx intervention during existing, multilevel church activities using a culturally-tailored COVID19 Tool Kit inclusive of digital tools consisting of: a) individual self-help materials and automated/tailored text messages; b) virtual supportive group seminars about COVID19; c) virtual/in-person church services with COVID19 related materials/activities (e.g., sermons, pastors modeling testing, testimonials, bulletins); and d) church-community level COVID19 testing and LTC services (e.g., healthcare, prevention programs, community resources, contact tracing) provided virtually by community health workers. All churches will host COVID19 testing events. First, a pilot study site will be used to test project feasibility followed by the 16 RCT faith-based study sites. Social, ethical, behavioral implications (SEBI) data will also be collected. All data will be made available to the Rapid Acceleration of Diagnostics Underserved Populations (RADxUP) Data Consortium.

Specific Aims (SA):

SA 1. Test a tailored TPB-guided multilevel, COVID19 intervention against a nontailored AC arm on uptake of COVID19 testing, and LTC/CTA & prevention behaviors with African American church-populations at 6 months.

Hypothesis: The tailored, TPB testing/LTC intervention will attain higher testing rates than AC at 6 months.

SA 2. Evaluate roles of potential mediators and moderators related to COVID19 testing among church-affiliated African Americans at 6 months to determine modifiable facilitators/barriers.

SA 3. Conduct a process evaluation to understand study implementation facilitators, barriers, and fidelity; and examine relationships between implementation, intervention dose and exposure, and intervention outcomes to identify and improve essential intervention components.

Significance: This novel study is the first to fully test a COVID19 testing and LTC intervention in African American churches. It could provide a theory-based, multilevel model for delivering scalable, wide-reaching COVID19 testing and LTC by supporting African American faith leaders with culturally-appropriate, easy-to-use tools and health agency partnerships. It could have a major impact on uptake of COVID19 testing, inform on LTC and contact tracing, and streamline future vaccine delivery in African American communities hard hit by COVID19.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be eligible to participate if they are: a) self-identified as African American/Black; b) aged 18 or older; c) willing to participate in 2 surveys after church services, electronically, by phone, or in the study's office space; d) willing to provide contact information (i.e., two phone numbers, mailing/email address, phone numbers for two persons with whom they have ongoing contact; and e) regularly attend church (>once a month) or use church outreach services (e.g., daycare services, food programs) > 4 times/year. Exclusion criteria include: persons with plans to move from KC metro area over the next 12 months and non-English speaking/reading persons.

Exclusion Criteria:

* Living outside of the Kansas or Missouri geographical areas

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1013 (Actual)
Dates: Start 2021-06-06 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
COVID-19 testing uptake | Change from baseline at 6 months
  COVID19 Testing will be assessed via self-report (ever, last 6 months, month/day/year) and objectively assessed with data reports provided by the Kansas City MO Health Department

SECONDARY OUTCOMES:
Linkage to care | Change from baseline at 6 months
  Utilization of linkage to care services via self-report (types of services received, number of contacts, engagement in contact tracing) and objectively assessed with data reports provided by the Kansas City MO Health Department
COVID-19 prevention behaviors | Change from baseline at 6 months
  Engagement in COVID19 prevention/mitigation behaviors (eg, mask wearing, 6 ft social distancing, hand washing, sheltering in place/quarantine)

CONTACTS AND LOCATIONS:
Overall Officials: Jannette Berkley-Patton, PhD, Principal Investigator — UMKC School of Medicine
Locations (10):
- United States (10):
  - Rhema Church, Independence, Missouri
  - Boone Tabernacle, Kansas City, Missouri
  - Centennial United Methodist Church, Kansas City, Missouri
  - Kansas City Health Department, Kansas City, Missouri
  - University of Missouri-Kansas City, Kansas City, Missouri
  - Sunlight Missionary Baptist Church, Kansas City, Missouri
  - Apostolic Church of God, Kansas City, Missouri
  - Jameson Memorial Temple, Kansas City, Missouri
  - Kingdom Word Ministries, Kansas City, Missouri
  - Memorial Church International, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared per a data agreement plan with NIH and with Duke University as part of the Rapid Acceleration of Diagnostics Underserved Populations initiative. Additionally de-identified data can be requested directly from the primary and secondary contacts. We will make the de-identified data and associated documentation available to potential requesters only under a data sharing agreement (based on the requester's proposed use of the data and under the guidance of our Institutional Review Board) that provides for: (1) a commitment to using the data only for research purposes and to not identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.
Supporting Information: Study Protocol, ICF
Time Frame: March 2023